CLINICAL TRIAL: NCT00908427
Title: Impact of 80 Watt KTP Photoselective Laser Vaporization Prostatectomy on Severity of Obstruction in Benign Prostatic Hyperplasia: 6-Month Results of a Nonrandomized Prospective Trial
Brief Title: Impact of 80 W KTP Laser Vaporization Prostatectomy on Severity of Obstruction in Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sung Won Lee/Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-05-09
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2009-05

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia
Keywords: benign prostatic hyperplasia; KTP laser; transurethral resection of prostate; urinary bladder neck obstruction
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia; Urinary Bladder Neck Obstruction | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): PVP group
  Interventions: Procedure: photoselective vaporization prostatectomy (PVP)
- 2 (Active Comparator): TURP group
  Interventions: Procedure: Transurethral resection of the prostate

INTERVENTIONS:
Procedure: photoselective vaporization prostatectomy (PVP) — PVP using 80 W KTP laser with a Greenlight system (GreenLight PVTM, Laserscope®, San Jose, CA)
  Other Names: PVP
  Arms: 1
Procedure: Transurethral resection of the prostate — Standard transurethral resection of the prostate using electrocautery loop
  Other Names: TURP
  Arms: 2

SUMMARY:
The purpose of this study is to compared the efficacy of 80W KTP photoselective laser vaporization prostatectomy (PVP) and transurethral resection of the prostate (TURP) in reducing the volume of prostate and relieving the obstruction in men with benign prostatic hyperplasia (BPH) on non-randomized controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic BPH
* International Score Prostate Symptom (IPSS) of 13 or greater
* prostate volume of 30 to 100 ML
* Peak urinary flow rate (Qmax) less than 15 mL/s with a voided volume of >125 mL and a PVR <350mL
* Able to give fully informed consent

Exclusion Criteria:

* Subjects with histological diagnosis of prostate cancer
* Subjects with history of chronic urinary retention
* Subjects with urethral stricture,
* Subjects with bladder neck contracture
* Subjects with urinary tract infection
* Subjects with prostate volume on TRUS of >100 mL
* Subjects with suspected neurogenic bladder dysfunction
* Subjects who, in the opinion of investigator, are not likely to complete the study for whatever reason

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-06; Primary Completion 2006-05 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The changes of bladder outlet obstruction index (BOOI) | 6months

SECONDARY OUTCOMES:
The changes of Quality of Life (QoL) parameters | 6, 12 months
The changes of Uroflowmetry (UFM) and Postvoid residual urine(PVR) | 6, 12 months
The changes of detrusor pressure at maximum flow rate (PdetQmax)parameters | 6months
The changes of International Prostatic Symptom Scores (IPSS) | 6, 12 months
The changes of Schafer obstruction grade parameters | 6months
The changes of prostate volume | 6, 12 months
postoperative catheterization days | immediate postoperative period
Complications | During all study periods
The changes of the hemoglobin and the serum sodium and the serum PSA | immediate postoperative period
The change of IIEF score | 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Won Lee, Ph.D.,M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea